CLINICAL TRIAL: NCT03535428
Title: Venous Thrombo-embolic Complication prévention in Pelvic Surgery
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PREVENTION MTEVbassin
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-07

CONDITIONS: Venous Thromboembolism; Pelvic Surgery
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VENOUS exploration
  Interventions: Diagnostic Test: VENOUS exploration

INTERVENTIONS:
Diagnostic Test: VENOUS exploration — venous echo doppler ultrasound and abdo pelvic scanner in the 48h before surgery

SUMMARY:
Pelvic fracture surgery are very high thrombotic risk surgery with about 10% to 50% venous thrombo embolic complications and 0.5% to 10% of pulmonary embolism. The ST JOSEPH's Hospital have almost 60 cases per year . Following a fatal pulmonary embolism per operatory the team has set up a venous exploratory protocol before surgery.

This protocol includes a venous doppler ultrasound of lower limbs associated to a abdo pelvic scanner in the 48hours before surgery.

The aim is to evaluate this new protocol efficacy on prevention of thrombo embolic complications in pelvic fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* pelvic fracture with surgery indication
* age above 18 years

Exclusion Criteria:

* pelvic fracture without surgery indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with pelvic surgery indication consulting surgeons
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
major thrombo-embolic events | Day 10 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: BONHOMME Stéphanie, MD, Principal Investigator — GHPSJ; RIOUALLON Guillaume, MD, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France